CLINICAL TRIAL: NCT01269034
Title: New Onset Type 1 Diabetes: Role of Exenatide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-435; 3R01DK077166-05S1 (NIH)
Record Dates: First submitted 2010-12-29; First posted 2011-01-04 (Estimated); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes Milletus; diabetes; healthy controls; exenatide; byetta
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Exenatide; Insulin, Long-Acting; Insulin Aspart; Insulin Lispro; Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (4):
- Part A (Experimental): Exenatide and long acting insulin before the boost.
  Interventions: Drug: Exenatide
- Part B (Active Comparator): Rapid and long acting insulin before the boost
  Interventions: Drug: Rapid and long acting insulin
- Part C (Active Comparator): long acting insulin+ rapid acting+1.25 mcg Exenatide before the boost
  Interventions: Drug: long acting insulin + rapid acting + 1.25 mcg Exenatide
- Healthy controls (No Intervention): healthy controls without any medication before the boost.

INTERVENTIONS:
Drug: Exenatide — 1.25 mcg before the boost sub-cutaneously.
  Other Names: Byetta
  Arms: Part A
Drug: Rapid and long acting insulin — Depends on their Carbohydrate ratio and body needs
  Other Names: Novolog/ Humalog; Lantus/ Levemir
  Arms: Part B
Drug: long acting insulin + rapid acting + 1.25 mcg Exenatide — Depends on their body needs.
  Other Names: Lantus; Levemir
  Arms: Part C

SUMMARY:
There are many recent advances in insulin treatment of type 1 diabetes, however after a meal sugars are always a concern. There is a drug Exenatide (Byetta) which is FDA approved to treat people with type 2 diabetes which helps correct their glucoses (sugars) after meals. This study is going to test whether this drug can improve the after meal sugars in people with new onset type 1 diabetes. To test this you will be given a dose of exenatide (1.25 mcg) and long acting insulin or inulin alone before the boost. There is also a placebo group (healthy subjects) who do not get any medication before the boost. Insulin levels and other hormones that affect blood glucose as well as your sugar will be measured by a series of blood tests. The role exenatide as compared to insulin alone will be examined to prevent low blood sugars which might occur because of food staying longer in the stomach than usual or due to the suppression of a hormone called glucagon which increases blood sugar. If you qualify you will be given exenatide (Byetta 1.25 mcg) along with insulin or insulin alone. You and the researchers will not know which dose you are taking at any single visit. A total of 20 people in which some will be children aged 12- 18 years will participate, being diagnosed within 3 months of having been found to have type 1 diabetes.

DETAILED DESCRIPTION:
The specific aims of this study are to determine the following:

1. The role of exenatide as compared to insulin monotherapy in reducing postprandial hyperglycemia.
2. The role of exenatide on postprandial glucagon and gastric emptying.
3. The effect of long acting insulin on postprandial glucose excursions, glucagon concentrations and gastric emptying.
4. Postprandial glucose excursions, glucagon concentrations and gastric emptying in normal healthy controls.

Study Design:

A randomized, non-blinded trial with a crossover design will be used. Following informed consent and with appropriate subject assent, all subjects will have a screening visit. Following the screening visit, subjects with T1DM will undergo 3 studies: Part A (exenatide and long acting insulin), Part B (rapid and long acting insulin) and Part C (long acting insulin only). The subjects will be admitted to the CRC on three separate occasions, at least 3-4 weeks apart. The three studies will be performed in a random order and the randomization will be done using a computerized system. The healthy controls will undergo a single study visit. Except for the absence of diabetes, the healthy controls will be identical to the study subjects. Subjects with new onset diabetes will be compared to healthy controls.

During the study, if blood glucose values in a subject are less than 55 mg/dl, IV glucose of 5-15 grams will be administered to achieve euglycemia (90-130 mg/dl). 1-2 doses of IV glucose should correct hypoglycemia. If more than 3 doses are required to achieve euglycemia, the study will be terminated, the subject will be offered a meal tray and blood sugar rechecked to ensure euglycemia. If blood sugar at any time is more than 350 with moderate ketones, the study will be terminated.

At around 1 PM (270 min), lunch will be provided (consistent carbohydrate meal) and insulin will be given as per the subject's prescribed regimen. The subject will be discharged home with a designated driver due to the risk of hypoglycemia.

A subject will be withdrawn from participating in the study if he/she meets any of the following conditions: 1)develops a chronic disease 2)develops anemia 3)becomes pregnant 4)develops a weight loss of greater than 10 pounds for unspecified reasons 5)loss of contact- if the investigators are unable to reach a study subject (within 2 months of screening or completion of the first study) by phone or mail to schedule the next appointment. All study subjects (that are withdrawn from the study) will receive a phone call and a letter notifying them that they have been withdrawn.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 12-18 years of age at the time of enrollment.
2. Diagnosed with antibody positive T1DM in the past 3 months.
3. Otherwise healthy except for their TIDM and treated hypothyroidism.
4. Females must have a negative pregnancy test.
5. Hemoglobin equal to or greater than 12 g/dl before each study.
6. Weight greater than 44 kg.

Exclusion Criteria:

1. Any chronic disease: leukemia, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis etc, except for diabetes and hypothyroidism.
2. Any medications that may affect glucose metabolism.
3. Abnormal AST, ALT, amylase, lipase, creatinine (more than 3 times normal values).
4. Lack of a supportive family environment as detected by the clinicians and/or social workers.
5. History of substance abuse (evaluated by medical history and CRAFFT questionnaire which will be administered at the screening visit).
6. Positive pregnancy test in females.
7. Lactating and nursing mothers.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjitha Katikaneni, MB; BS, Study Director — Montefiore Children's hospital
Locations (1):
- Albert Einstein CRC- West Campus, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 people in which some will be children aged 12- 18 years will participate, being diagnosed within 3 months of having been found to have type 1 diabetes.
Pre-assignment Details: "Each participant only received one part (A,B, or C) and did not cross over to the subsequent parts
Period: Overall Study
Arm/Group | Part A | Part B | Part C | Healthy Controls
Started | 1 | 2 | 1 | 9
Completed | 0 | 2 | 1 | 9
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data for this outcome measure are no longer accessible; the PI has left institution and all efforts to locate the data have been exhausted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Part C | Healthy Controls | Total
Number analyzed (Participants) | 1 | 2 | 1 | 9 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 6 | 8
  Between 18 and 65 years | 1 | 1 | 0 | 3 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 5 | 7
  Male | 0 | 1 | 1 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 5 | 7
  Not Hispanic or Latino | 0 | 1 | 1 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 1 | 8 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Role of Exenatide as Compared to Insulin Monotherapy in Reducing Postprandial Hyperglycemia.
Description: Data for this outcome measure are no longer accessible; the PI has left institution and all efforts to locate the data have been exhausted.
Time Frame: February 2013
Population: The original PI and their entire team left the institution. Despite repeated efforts to contact the PI and study team members, the PI and study team members refused to disclose any collected data. Additionally, no secondary information sources such as study publications exist from which to summarize collected data
Arm/Group | Part A | Part B | Part C | Healthy Controls
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: The Role of Exenatide on Postprandial Glucagon and Gastric Emptying.
Description: as for outcome 1
Time Frame: February 2013
Population: as for outcome 1
Arm/Group | Part A | Part B | Part C | Healthy Controls
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Postprandial Glucose Excursions, Glucagon Concentrations and Gastric Emptying in Normal Healthy Controls.
Description: as for outcome 1
Time Frame: February 2013
Population: as for outcome 1
Arm/Group | Part A | Part B | Part C | Healthy Controls
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 years
Description: While Adverse Events were monitored/assessed, none were observed
Arm/Group | Part A | Part B | Part C | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/1 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/1 | 0/9
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/1 | 0/9

LIMITATIONS AND CAVEATS:
The original PI and their entire team has left the institution. Repeated attempts for complete data have gone unanswered. Outcome measure data is not available to provide full and complete results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-04-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT01269034/Prot_000.pdf